CLINICAL TRIAL: NCT00557752
Title: Non-Invasive Ventilation in Early Severe Posttraumatic Hypoxia: a Randomized Controlled Trial
Brief Title: Efficacy of Non-Invasive Mechanical Ventilation in Early Hypoxia Secondary to Thoracic Trauma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Review Board stopped the study after interim analysis reaching stopping rule for efficacy.
Sponsor: Hospital Virgen de la Salud (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Ramon Galvez Zaloña, SESCAM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06001-00
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Post-Traumatic Respiratory Failure
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Addition to the standard therapy of non-invasive mechanical ventilation. Continuously for the first 24 hours, then trials to discontinuation every 24 hours. Interface adjusted for the associated injuries.
  Interventions: Device: Non-invasive ventilation
- 2 (No Intervention): Standard therapy for severe post-traumatic hypoxia: pain control with epidural anesthesia and oxygen.

INTERVENTIONS:
Device: Non-invasive ventilation — Applied continuously for the first 24 hours, then every 24 hours, trial of discontinuation. Interface specific for the associated injuries.
  Arms: 1

SUMMARY:
* Severe post-traumatic hypoxia is mainly due to lung contusion. The intubation rate of these patients is near 20%.
* Treatment before intubation is needed, is based on pain control with epidural anesthesia and oxygen.
* The investigators' hypothesis is that adding non-invasive mechanical ventilation to the standard treatment can reduce the intubation rate if applied early in the course of the disease.
* As thoracic trauma is often associated with injuries in other body regions that may increase the complications of the technique, specific contraindications have been described.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Informed consent obtained.
* pO2/FiO2 <200 for more than 8 consecutive hours in the first 48 hours after thoracic trauma.

Exclusion Criteria:

* Orotracheal intubation indicated for any other reason.
* Standard contraindication for non-invasive ventilation (active gastro-intestinal haemorrhage, low level of consciousness, multiorgan failure, airway control problems, lack of cooperation, hemodynamic instability).
* Severe traumatic brain injury.
* Facial trauma with pneumocephalus, skull base fracture, orbit base fracture, any facial fracture involving a sinus.
* Cervical injury with specific treatment contraindicating a facial mask.
* Bronco-pleural fistula.
* Gastro-intestinal trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Intubation rate | 1 month

SECONDARY OUTCOMES:
Pneumothorax rate | 1 month
Pneumonia rate | 1 month
Intensive Care Unit stay | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Hernandez, Dr., Principal Investigator — Hospital Virgen de la Salud
Locations (2):
- Spain (2):
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Virgen de la Salud, Toledo, Toledo

REFERENCES:
- [Result] British Thoracic Society Standards of Care Committee. Non-invasive ventilation in acute respiratory failure. Thorax. 2002 Mar;57(3):192-211. doi: 10.1136/thorax.57.3.192. No abstract available. PMID 11867822
- [Derived] Hernandez G, Fernandez R, Lopez-Reina P, Cuena R, Pedrosa A, Ortiz R, Hiradier P. Noninvasive ventilation reduces intubation in chest trauma-related hypoxemia: a randomized clinical trial. Chest. 2010 Jan;137(1):74-80. doi: 10.1378/chest.09-1114. Epub 2009 Sep 11. PMID 19749006